CLINICAL TRIAL: NCT02060071
Title: Endothelial Progenitors in Aortic Stenosis: Association With Aortic Stenosis Progression, Severity, Symptoms and Left Ventricular Function Assessed by 2D Strain Echocardiography
Brief Title: Endothelial Progenitors in Aortic Stenosis: Association With Aortic Stenosis Progression and Severity
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaplan Medical Center (Other)
Responsible Party: Principal Investigator, Sara Shimoni, MD, Director of non Invasive Cardiology Unit, Kaplan Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: kap118711ctil
Record Dates: First submitted 2014-02-03; First posted 2014-02-11 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-02

CONDITIONS: Aortic Stenosis; Cardiac Death
Keywords: aortic stenosis
MeSH Terms: conditions — Aortic Valve Stenosis; Death | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aortic setnsosi (Other): blood test
  Interventions: Other: Blood test
- controls (Other): blood test
  Interventions: Other: Blood test

INTERVENTIONS:
Other: Blood test — Blood test

SUMMARY:
There is a correlation between endothelial progenitor cells (stem cells) and stenosis of the aortic valve.

DETAILED DESCRIPTION:
Degenerative aortic valve (AV) stenosis (AS) is the most common valvular disease and increases in prevalence with age. Severe aortic valve stenosis accounts for considerable disease and death, especially in older patients. Aortic valve stenosis is the primary indication for valve replacement in western countries, and the number will only increase as elderly people are a growing subpopulation. Measures to identify AV disease earlier, to identify factors that influence disease progression and treat AV disease pharmacologically or with less invasive approaches would be a significant improvement over the current standard of care. These advances will only be possible with a better understanding the mechanisms underlying valve development and disease. Preliminary data suggest a novel pathophysiological concept for impaired valvular endothelial cells regeneration, leading to the progression of age-associated calcific AV disease and a potential treatment target is the disrupted endothelial cell layer of the valve leaflet.

The research objectives are:

1. To assess the number and function of endothelial progenitor cellss and apoptotic endothelial progenitor cellss in patients with mild, moderate and severe aortic stenosis.
2. To study the association between aortic stenosis progression, severity, symptoms and left ventricular function and the number and function of circulating endothelia progenitor cells. By understanding the correlation between valve severity, left ventricular longitudinal function and endothelial progenitor cells we will indentify high risk patients population that need early intervention. We hope to add new information on the pathogenesis of aortic stenosis and to indentify factors that predict disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Aortic stenosis
* Control with aortic stenosis

Exclusion Criteria:

* No

Ages: 18 Years to 92 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-07; Primary Completion 2014-02 (Actual); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Cardiac death or need for intervantion in correlation to endothelial progenitor cells | 4 years
  We will assess wether endothelial progenitor cells can predict outcome

CONTACTS AND LOCATIONS:
Overall Officials: Sara Shimoni, MD, Principal Investigator — Kaplan Medical
Locations (1):
- Kaplan Medical Center, Rehovot, Israel